CLINICAL TRIAL: NCT04530994
Title: A Maralixibat Expanded Access Program for Patients With Cholestatic Pruritus Associated With Alagille Syndrome
Brief Title: A Maralixibat Expanded Access Program for Patients With Cholestatic Pruritus Associated With Alagille Syndrome (ALGS)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Collaborators: Clinigen, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MRX-EAP
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Alagille Syndrome
Keywords: Liver Disease; ALGS; Maralixibat; Bile Duct Diseases; Digestive System Diseases; Biliary Tract Diseases; Cholestasis; Pruritis
MeSH Terms: conditions — Alagille Syndrome; Liver Diseases; Bile Duct Diseases; Digestive System Diseases; Biliary Tract Diseases; Cholestasis; Pruritus | interventions — maralixibat

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: maralixibat — Maralixibat is an Apical Sodium-dependent Bile acid Transporter (ASBT) inhibitor

SUMMARY:
An open-label, single-arm, multi-centre program providing treatment access to ALGS patients with cholestatic pruritus in the US. Access can be requested through Clinigen Healthcare Ltd via email MirumALGS@clinigengroup.com or telephone +1-877-768-4303.

DETAILED DESCRIPTION:
The objective of this EAP is to provide access to maralixibat for eligible ALGS patients with cholestatic pruritus. Participants will be treated with 400 µg/kg/day with safety and tolerability evaluated on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent and assent provided, as applicable, per Institutional Review Board (IRB) or Ethics Committee (EC)
2. Clinical and/or genetic diagnosis of ALGS
3. Male or female participants aged >12 months and ≥5 kg with clinically significant cholestatic pruritus associated with ALGS
4. Willingness to adhere to an acceptable method of contraception until treatment discontinuation by females of childbearing potential who are sexually active or who become sexually active during the program
5. No other therapeutic options or access to any ongoing ALGS clinical trials

Exclusion Criteria:

1. Diagnosis with a cholestatic liver disease other than ALGS
2. Female who is pregnant or breastfeeding
3. Clinically significant cardiovascular, hepatic, gastro-intestinal, pulmonary, neurologic, infectious or renal disease or other medical condition that, in the opinion of the physician or Medical Monitor, would preclude participation in the program
4. Past medical history of compensated or decompensated cirrhosis
5. Presence of any other disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of maralixibat or its mode of action

Min Age: 12 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - University of California San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Advent Health, Orlando, Florida
  - Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Hospital at Montefiore, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Genetics Home Reference - Alagille syndrome — https://ghr.nlm.nih.gov/condition/alagille-syndrome
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com
- See also: Mirum webpage specific to ALGS EAP — https://algseap.com/